CLINICAL TRIAL: NCT03825211
Title: Continuous Versus Discontinuous Suture in the Perineals Lesions Produced During Delivery in Primiparous: Maternal Results: A Randomized Controlled Trial
Brief Title: Continuous Versus Discontinuous Suture in the Perineals Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Juan Miguel Martinez-Galiano, Principal Investigator, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Ujaen Sutura Lesiones
Record Dates: First submitted 2019-01-25; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Perineal Tear; Episiotomy Wound

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous suture (Experimental): All parts of the perineal lesion (vaginal mucosa , perineal muscle and skin) be sutured with the same suture thread. A single suture for perineal lesion
  Interventions: Procedure: Continuous suture in the perineals lesions
- Discontinuous suture (Active Comparator): Interrupted suture technique: vaginal mucosa, perineal muscle and skin are sutured with separate and different threads, that is, the vaginal mucosa is sutured with a thread, then independently the perineal muscle is sutured with another type of thread and finally the skin is also sutured independently with another different thread. Three independent sutures for each of the parts that form a single perineal lesion
  Interventions: Procedure: Discontinuous suture in the perineals lesions

INTERVENTIONS:
Procedure: Continuous suture in the perineals lesions — A continuous suture of the vagina, muscle and skin is performed continuously, without knotting or cutting the suture thread.
  Arms: Continuous suture
Procedure: Discontinuous suture in the perineals lesions — Suture the muscle independently of the vagina and independently of the skin
  Arms: Discontinuous suture

SUMMARY:
The hypothesis: Women who have a continuous suture have better health outcomes Two types of sutures were placed in the perineal lesion, using different techniques. Group A received continuous sutures and Group B had interrupted sutures placed. The women were followed-up as follows: Day of childbirth and in the postpartum period.

DETAILED DESCRIPTION:
The hypothesis: Women who have a continuous suture have better health outcomes Two types of sutures were placed in the perineal lesion, using different techniques. Group A received continuous sutures and Group B had interrupted sutures placed. The women were allocated to a treatment group using a computer-generated random numbers table. The sequence was placed in individual opaque envelopes that were opened when a woman met the inclusion criteria.

The health personnel that carry out the sutures had taken a training course on continuous suture technique and had at least one year experience in this technique. Additionally, this person had a minimum of five years of experience in attending deliveries and therefore also in the suturing of perineal lesions. The sutures were placed by ten trained midwives. Around 5% of the midwives in Torrecardenas, 10% in the Hospital Complex of Jaen, 12% in Granada, and 20% of the midwives in Ubeda and Linares participated.

Data collection Data was collected on sociodemographic variables, type of perineal trauma (tear of second-degree or episiotomy), type of suture used, time spent placing suture, number of suture packets used, complications, analogical scale of pain, type of pain, need for analgesia, wound condition, care performed, urinary and/or fecal incontinence, start of sexual relations, start of physical activity and type of newborn feeding. It was also collected the start and type of delivery, medication during dilation, type of analgesia used, gestational week, duration of dilation, second stage labor and delivery, and data on the newborn.

Information was gathered by midwives which interviewed the women in the labor room, providing them with an informed consent form, and hiding the suture technique that was going to be used. The rest of the data were obtained from the clinical history, maternal record book and phone calls made for the follow-up. The women did not know at any point which suture technique had been used.

Follow-up

The women were followed-up as follows:

Day of childbirth: in the postpartum period, the midwife collected data on the type of delivery, need for epidural analgesia, duration of dilation, stage two of labor, delivery, type of perineal trauma, time used to place suture, number of suture packets, wound complications, newborn weight and the Apgar score at one minute and at five minutes. After the suture was placed, they assessed pain on the pain scale and assessed the wound.

Follow-up after delivery was done at two hours, 24 hours, 15 days and three months. Pain, need for analgesia, wound condition, sphincter incontinence and the start of sexual relations were assessed (15 days and three months).

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Primiparous
* Singleton and eutocic delivery
* Second-degree perineal tear or an episiotomy as part of labor
* Newborn weight between 2500 g and 4000 g

Exclusion Criteria:

* Language barrier (to no speak spanish)
* Problems related to the pelvic floor prior to labor (prolapse, incontinence, vulva varices)
* Dyspareunia or sexual dysfunction
* Hemorrhoids perceived as uncomfortable or painful

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Analogical scale of pain | After delivery was done at two hours
  It consists of a line horizontal 10 centimeters, at the ends of which are the extreme expressions of a symptom In the left is the absence or less intensity and in the right the greater intensity
Numerical verbal scale for pain | After delivery was done at 24 hours
  Scale numbered 1-10, where 0 is the absence and 10 the highest intensity, the patient selects the number that best assesses the intensity of the symptom.
Numerical verbal scale for pain | After delivery was done at 15 days
  Scale numbered 1-10, where 0 is the absence and 10 the highest intensity, the patient selects the number that best assesses the intensity of the symptom.
Numerical verbal scale for pain | After delivery was done at three months.
  Scale numbered 1-10, where 0 is the absence and 10 the highest intensity, the patient selects the number that best assesses the intensity of the symptom.

SECONDARY OUTCOMES:
Questionnaire | After delivery was done 15 days
  The woman was asked if she had involuntary urine losses.The possible answer is "yes" (she has incontinence) or "no" (she has no incontinence)
Questionnaire | After delivery was done three months.
  The woman was asked if she had involuntary urine losses. The possible answer is "yes" (she has incontinence) or "no" (she has no incontinence)
Questionnaire on Women Sexual Function (WSF) | After delivery was done at three months.
  This questionnaire has been validated in Spain. The instrument is composed of two types of domains: the evaluators of sexual activity, which are answered by a Likert scale of five values; and the descriptive ones, which have no quantitative value and help to know issues such as the frequency of sexual activity or the existence of sexual dysfunction in the respondent. It consists of 14 items, an alternative item and a question to open the questionnaire. To diagnose sexual dysfunction, only 6 questions are counted: Desire, Excitement, Lubrication, Orgasm, Problems with vaginal penetration, Anticipatory anxiety. Diagnostic results are categorized into: severe, moderate and no-disorder disorder. It does not establish degrees of dysfunctionality of sexual function, it is not shown in validation study if there is a cutoff point. The maximum score of this questionnaire is 100, which is interpreted as "without sexual dysfunction".

REFERENCES:
- [Derived] Martinez-Galiano JM, Arredondo-Lopez B, Hidalgo-Ruiz M, Narvaez-Traverso A, Lopez-Moron I, Delgado-Rodriguez M. Suture type used for perineal injury repair and sexual function: a randomised controlled trial. Sci Rep. 2020 Jun 29;10(1):10553. doi: 10.1038/s41598-020-67659-2. PMID 32601329
- [Derived] Martinez-Galiano JM, Arredondo-Lopez B, Molina-Garcia L, Camara-Jurado AM, Cocera-Ruiz E, Rodriguez-Delgado M. Continuous versus discontinuous suture in perineal injuries produced during delivery in primiparous women: a randomized controlled trial. BMC Pregnancy Childbirth. 2019 Dec 16;19(1):499. doi: 10.1186/s12884-019-2655-2. PMID 31842788